CLINICAL TRIAL: NCT04249323
Title: A Phase 1 Adaptive Dose, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Orally Administered CORT113176 in Healthy Subjects, With an Optional Pharmacological Effects Cohort
Brief Title: Single and Multiple Ascending Dose Study of CORT113176 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CORT113176-650; 2019-004258-27 (EudraCT Number)
Record Dates: First submitted 2020-01-29; First posted 2020-01-30 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Dosage Forms; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1: SAD Cohorts A through H CORT113176 (Experimental): Cohorts will receive a single dose of CORT113176 lipid capsule formulation by mouth on Day 1 in a fasted or fed state. Cohort A will receive a 50-mg dose in a fasted state. Cohort B will receive a ≤3-fold increase in dose from Cohort A in a fasted state; the dose will be determined after evaluation of safety and PK data for Cohort A. Subsequent cohorts will receive a ≤3-fold increase in CORT113176 dose from the previous cohort in a fasted or fed state; the dose and prandial state will be determined after evaluation of safety and PK data from previous cohorts. Following interim review of PK data, an alternative lipidic formulation may be administered beginning with Cohort B.
  Interventions: Drug: CORT113176 Lipid Capsule Formulation
- Part 1: SAD Cohorts A through H Placebo (Placebo Comparator): Cohorts will receive a single dose of placebo matching CORT113176 lipid capsule formulation by mouth on Day 1. The dose of placebo, prandial state, and choice of formulation will match that used for the corresponding SAD cohorts receiving CORT113176.
  Interventions: Drug: Placebo matching CORT113176 Lipid Capsule Formulation
- Part 2: MAD Cohorts A through D CORT113176 (Experimental): Cohorts will receive once- or twice-daily doses of CORT113176 lipid capsule formulation by mouth for 14 days. The anticipated exposure will not exceed the highest exposure considered safe and well-tolerated during Part 1. The dose schedule and prandial state will be determined after evaluation of safety and PK data from Part 1. The choice of formulation of CORT113176 to be used in Part 2 will depend on data review for Part 1.
  Interventions: Drug: CORT113176 Lipid Capsule Formulation
- Part 2: MAD Cohorts A through D Placebo (Placebo Comparator): Cohorts will receive once- or twice-daily doses of placebo matching CORT113176 lipid capsule formulation by mouth for 14 days. The dose of placebo, prandial state, and choice of formulation will match that used for the corresponding MAD cohorts receiving CORT113176.
  Interventions: Drug: Placebo matching CORT113176 Lipid Capsule Formulation
- Part 3: Single Dose Pharmacodynamic Effect (Experimental): In Period 1, participants will receive a single dose of prednisone 25 mg tablet by mouth on Day 1 in a fasted or fed state. After a 7-day washout, in Period 2, participants will receive a single dose of prednisone as in Period 1 plus a single dose of CORT113176 lipid capsule formulation by mouth on Day 1 in a fasted or fed state. The dose of CORT113176 and the prandial state will be determined after evaluation of safety and PK data from Part 1. The choice of formulation of CORT113176 to be used in Part 3 will depend on data review for Part 1. Part 3 will proceed only if sufficiently high plasma CORT113176 exposure is achieved in Part 1.
  Interventions: Drug: CORT113176 Lipid Capsule Formulation; Drug: Prednisone

INTERVENTIONS:
Drug: CORT113176 Lipid Capsule Formulation — CORT113176 Lipid Capsule Formulation 10-200 mg for oral administration
  Arms: Part 1: SAD Cohorts A through H CORT113176; Part 2: MAD Cohorts A through D CORT113176; Part 3: Single Dose Pharmacodynamic Effect
Drug: Placebo matching CORT113176 Lipid Capsule Formulation — Placebo matching CORT113176 Lipid Capsule Formulation 10-200 mg for oral administration
  Arms: Part 1: SAD Cohorts A through H Placebo; Part 2: MAD Cohorts A through D Placebo
Drug: Prednisone — Prednisone standard release tablets 1 x 20 mg plus 1 x 5 mg for oral administration
  Arms: Part 3: Single Dose Pharmacodynamic Effect

SUMMARY:
This is a 3-part, first-in-human study of single ascending doses (SAD; Part 1) and multiple ascending doses (MAD; Part 2) of CORT113176 in healthy participants; Part 3 is an optional part to investigate whether CORT113176 ameliorates the effects of prednisone on various pharmacodynamic (PD) endpoints. The 3 parts may not be conducted entirely sequentially provided that this is justified by pharmacokinetic (PK) and safety data obtained from completed cohorts. The first MAD cohort will not start until data are available from at least 2 SAD levels to allow MAD administration in the fasted state, or until after a food-effect cohort has been dosed in the SAD phase to allow MAD administration in the fed state. The expected exposure for the daily MAD level at steady state (taking into consideration potential accumulation on repeat dosing) must not exceed the highest exposure considered to be safe and well tolerated during preceding SAD cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18.0 to 30.0 kg/m^2, inclusive
* Body weight ≤102 kg
* Willing to consume a high-fat breakfast, including pork
* Agrees to adhere to the contraception requirements of the protocol
* Additional criteria apply.

Exclusion Criteria:

* Received any investigational drug or device in a clinical research study within the last 90 days
* History of any drug or alcohol abuse in the last 2 years; a confirmed positive drugs of abuse test result
* Regular alcohol consumption; a confirmed positive alcohol breath test at screening
* Current smoker; a confirmed positive breath carbon monoxide reading; current user of e-cigarettes or nicotine replacement products in the last 6 months
* Female of childbearing potential, pregnant or breastfeeding
* Have a pregnant partner
* Clinically significant abnormal clinical chemistry, hematology, or urinalysis result
* Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV)
* Active renal or hepatic disease
* History of clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, respiratory, gastrointestinal, neurological, or psychiatric disorder
* Any form of cancer in the last 5 years (exceptions apply)
* History of adrenal insufficiency
* Have a condition that could be aggravated by glucocorticoid and/or mineralocorticoid blockade
* Currently using glucocorticoids or a history of systemic glucocorticoid use in the last 12 months or 3 months for inhaled products
* Additional criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Events | Part 1 SAD Cohorts: up to Day 9; Part 2 MAD Cohorts: up to Day 23; Part 3 Cohort: up to Day 19

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of CORT113176 | Before dosing and at pre-specified time points up to Day 9 (Part 1 SAD Cohorts), up to Day 23 (Part 2 MAD Cohorts), or Days 10-19 (Part 3 Cohort)
Time of Cmax (Tmax) of CORT113176 | Before dosing and at pre-specified time points up to Day 9 (Part 1 SAD Cohorts), up to Day 23 (Part 2 MAD Cohorts), or Days 10-19 (Part 3 Cohort)
Apparent Elimination Half-life (t1/2) of Plasma CORT113176 | Before dosing and at pre-specified time points up to Day 9 (Part 1 SAD Cohorts), up to Day 23 (Part 2 MAD Cohorts), or Days 10-19 (Part 3 Cohort)
Area Under the Plasma Concentration-time Curve (AUC) of CORT113176 | Before dosing and at pre-specified time points up to Day 9 (Part 1 SAD Cohorts), up to Day 23 (Part 2 MAD Cohorts), or Days 10-19 (Part 3 Cohort)
Serum Cortisol | Predose on Days 1 and 14 (Part 2 MAD Cohorts)
Serum Adrenocorticotropic Hormone (ACTH) | Predose on Days 1 and 14 (Part 2 MAD Cohorts)

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChb, BAO, MRCS, MFPM, Principal Investigator — Quotient Sciences
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided